CLINICAL TRIAL: NCT04790955
Title: Effect of Radiotherapy Concurrent With PARP Inhibitor + Temozolomide Combined With Immune Checkpoint Inhibitor on SCLC After Initial Treatment Failure
Brief Title: Effect of Combination Therapy on SCLC After Initial Treatment Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020IIT037
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Small-cell Lung Cancer
Keywords: SBRT, low dose radiotherapy, PARP inhibitor, PD-1,PD-L1
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SCLC patients after initial treatment failure are treated with SBRT and low-dose radiotherapy concurrent with PARP inhibitors + temozolomide +PD-1/PD-L1 inhibitors for two cycles at least, then PARP inhibitors+temozolomide+PD-1/PD-L1 inhibitors two cycles, PD-1/PD-L1 inhibitors maintenance therapy lasted for up to 2 years.

DETAILED DESCRIPTION:
SCLC is easy to relapse and drug resistance soon after initial treatment , although radiotherapy and chemotherapy is sensitive at first treatment. Topotecan monotherapy is recommended in the NCCN guidelines for second-line standard treatment and the CSCO SCLC guidelines for diagnosis and treatment 2020 edition, but its effective rate is low, 24% for platinum-sensitive relapse, 2-6% for platinum-resistant, overall PFS is about 3-4 months and OS is about 6-8 months. Although immunotherapy have been successful at the first-line and third-line treatments of SCLC in the extensive stage , the second-line treatment has not achieved a breakthrough, and the effective rate of third-line immune single drug is between 10-20%.It is an important challenge and breakthrough to effectively improve the efficacy and survival of second-line treatment of SCLC. Immunocombination therapy is an important strategy to improve the efficacy. Some studies have shown that PARP inhibitors and low-dose radiotherapy can improve the efficacy of immunotherapy. PARP inhibitors are not only sensitizers of chemoradiotherapy, but also immunomodulators. High dose radiotherapy has the effect of in situ vaccine and increases tumor antigen release presentation. Low dose radiotherapy promotes the penetration of immune cells into tumor stroma and tumor bed and increases immune response. The combination of high and low dose radiotherapy and immunization can improve the immune effect and increase the incidence of distant effect. So the objective of this study is to observe the efficacy and safety of second-line treatment of SCLC with SBRT and low-dose radiotherapy combined with PARP inhibitor + temozolomide and PD-1 /PD-L1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years old, ≤80 years old, expected survival ≥3 months;Pathologically confirmed SCLC with recurrence and metastasis after initial treatment;KPS score ≥70 points;Satisfied the following laboratory diagnostic indicators: hemoglobin ≥110g/L, leukocyte 4.0-10.0×109/L, neutrophils 2.0-7.5×109/L, platelet ≥100×109/L;Creatinine ≤ upper normal limit (UNL);ALT and AST≤2.5×UNL, alkaline phosphatase (ALP) ≤5×UNL, total bilirubin (TBIL) ≤ UNL;Signed informed consent.

-

Exclusion Criteria:

1. Pregnant or lactating women;
2. Secondary tumor;
3. HIV carriers;
4. Serious medical diseases such as heart and lung;
5. Patients with uncontrollable mental history, unable to cooperate with treatment;
6. Autoimmune system disease, symptomatic interstitial lung disease;
7. Patients with active infection, chronic infection, acute infection, etc., and body inflammation;
8. Patients who had used hormones or antibiotics 1 month prior to treatment. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SCLC patients after initial treatment failure
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
3 Month Objective Remission Rate | Up to 5 years
  The patients have complete remission and partial remission on 3 months after radiotherapy and chemotherapy.
Progression-Free Survival | From chemotherapy completion until progress or death, assessed up to 5 years
  Will be described using standard Kaplan-Meier methodologies. The median PFS time, 1-year rate, 3-year PFS rate and 5-year PFS rate will be estimated and presented with 90% confidence intervals.
Time To Progression | Up to 5 years
  Time involved from research start until progress for tumor

SECONDARY OUTCOMES:
Overall Survival | From chemotherapy completion until death, assessed up to 5 years
  Will be described using standard Kaplan-Meier methodologies. The median survival time, 1-year survival rate, 3-year survival rate , 5-year survival rate and will be estimated and presented with 90% confidence intervals.
Number of Participants With Serious Adverse Events Related to treatment | up to 5 years
  Toxicity assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4

CONTACTS AND LOCATIONS:
Overall Officials: Daxin Zhang, Dr., Study Director — First Affiliated Hospital of Harbin Medical University

IPD SHARING:
Plan to Share IPD: Undecided
There is not decision to make individual participant data available to other researchers